CLINICAL TRIAL: NCT06032221
Title: A Feasibility Study Assessing the Impact of At-home Infrared Temperature Monitoring (AITM) With Telemedicine Support in the Management of Patients With Potential for Diabetes Foot Ulceration
Brief Title: Study to Determine the Feasibility of Using an At-home Foot Temperature Monitoring Device (Thermidas)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays in device modifications. Unable to complete within MHRA timescale
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Robertson Centre for Biostatistics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: INGN21DI185
Record Dates: First submitted 2023-08-22; First posted 2023-09-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-02

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The purpose of the study is to determine if the Thermidas camera with telemedicine app is a feasible device in the 2 patient cohorts (15 patients who have had previous diabetes foot ulceration and 15 patients who are deemed to be high risk of foot ulceration)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- device feasibility (Other): All participants issued with Thermidas device
  Interventions: Device: Thermidas Vista Telehealth App

INTERVENTIONS:
Device: Thermidas Vista Telehealth App — Thermal camera with telemedicine app

SUMMARY:
This is a feasibility study, designed to assess the acceptability of At Home Temperature Monitoring (AITM) by patients at high risk of diabetes foot ulceration. The investigation hopes to identify any problems with the study design before progressing to a full-scale evaluation, and will assess the ease of use of the technology and if there are any barriers to using this.

Participants will be provided with an infrared camera and SMART phone and trained in how to use them. The participants will then be expected to capture images of both the plantar and dorsal aspects of their feet that will be sent to the research team for review. The two images will be captured once per day. The Intervention period will be 12 weeks.

If a raised temperature is identified, the participant will be offered a face to face review appointment where they will receive podiatry treatment (if required), ulcer prevention advice and more detailed thermal imaging. Patient and health care professional (HCP) questionnaires will be used at the start and end of the study period to assess quality of life impact and device ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or Female >/ = 18 years of age
* Diabetes Mellitus type 1 or 2 according to WHO criteria
* independently ambulatory
* deemed high risk/ in remission via SCI diabetes foot risk stratification tool
* expected to comply with study schedule

Exclusion Criteria:

* active foot ulcer or open amputation site
* active Charcot Neuro-osteoarthropathy
* active foot infection based on PEDIS classification criteria
* amputation proximal to the Chopart joint in one or both feet
* critical limb ischaemia (according to PEDIS classification)
* severe illness that would make 6-month survival unlikely based on the clinical judgement of the physician or podiatrist
* concomitant severe physical or mental conditions that limit the ability to follow the instructions of the study, based on the clinical judgement of the physician or podiatrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Device Feasibility - Completion | 12 weeks
  Participants successful completion of 12 weeks (percentage of all subjects who were enrolled in the study with ≥70% considered successful target (21 patients). This will assess if usage of the device on a daily basis over a specific period of time is practical
Device Feasibility - Withdrawal | 12 weeks
  Participants withdrawal (Percentage of all subjects who were enrolled in the study ≤30% considered successful target). A low withdrawal rate will demonstrate that usage of the device is practical over the time period
Device Feasibility - Compliance | 12 weeks
  No submission of images - i.e. no image submissions for 7-consecutive days on 2-occasions, generating 2-alerts over 12 weeks (absolute number of 'no submission' alerts). A lack of compliance with the study protocol will demonstrate low feasibility for regular device usage
Device Feasibility - Safety | 12 weeks
  Incidence of Serious adverse events (SAEs) and Adverse device reactions (ADRs)
Device Feasibility - Quality of life (QoL) utilising EQ-5D-5L instrument | 12 weeks
  Patient completion of EQ-5D-5L health utility score to obtain a health utility score at Baseline and at Week 12 (target 80% completion).
  (The EQ-5D-5L descriptive system comprises the same five dimensions as the EQ-5D-3L (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), but each dimension now has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each)
Device Feasibility - Health Economics | 12 weeks
  Health care utilisation and costs. The podiatrists will keep a log of time spent checking images and additional appointments generated in response to alerts. Costs will be calculated using staff time x staff payment costs
Device Feasibility - Staff feedback on device use | 12 weeks
  A focus group meeting with podiatrists will be scheduled at the end of the participant data collection period to obtain qualitative data relating to device use.
Device Feasibility - Patient feedback on device use | 12 weeks
  Patient completion of User Questionnaire Form (Week 12) (target 80% completion)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No